CLINICAL TRIAL: NCT02802202
Title: Validation of a Pressure Pain Threshold Scale in Patients Diagnosed With Myofascial Pain Syndrome and Fibromyalgia
Status: Completed | Type: Observational
Sponsor: California State University, Dominguez Hills (Other)
Responsible Party: Principal Investigator, Scott Cheatham, Assistant Professor (Division of Kinesiology), California State University, Dominguez Hills
Other Study IDs: #15-116
Record Dates: First submitted 2016-06-05; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Myofascial Pain Syndrome; Fibromyalgia
Keywords: Palpation; Chronic Pain; Muscle
MeSH Terms: conditions — Myofascial Pain Syndromes; Fibromyalgia; Chronic Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fibromyalgia: Individuals who met the criteria for a diagnosis of FM based upon the ACR diagnostic criteria.
- Myofascial Pain Syndrome: Individuals with a diagnosis of MPS that does not meet the American College of Rheumatology (ACR) diagnostic criteria for FM.
- Control: Individuals with no current or prior diagnosis consistent with MPS or FM.

SUMMARY:
To date, there are no valid and reliable pressure pain threshold scales for use in research or clinical practice. The existing manual palpation protocols and scales have limited support in the literature and our knowledge has not advanced since these scales were proposed in the 1990's. Therefore, the purpose of this investigation was to develop a valid and reliable PPTS in order to provide an objective means of assessing pressure pain thresholds and create a reliable method of communication among clinicians for individuals with a diagnoses characterized by MPS and FM. These conditions were chosen based on their high prevalence among chronic pain conditions and are also dependent upon the manual palpation examination for their diagnosis.

DETAILED DESCRIPTION:
The purpose of this investigation was to develop a valid and reliable PPTS in order to provide an objective means of assessing pressure pain threshold and to create a reliable method of communication among clinicians. Eighty-four participants (N=84) were enrolled in the study and assigned to three groups: FM (N=28), MPS (N=28), and control group (N=28). Participants were recruited from three sites. All participants were aged 18 to 65 years and met the inclusion criteria for 1 of the 3 groups. All participants were required to read, speak and write English as needed to complete forms and consent. The following criteria for each group was as follows:

1. Control group: Individuals with no current or prior diagnosis consistent with MPS or FM. No current injuries or integumentary abnormalities at the designated palpation sites.
2. MPS group: Individuals with a diagnosis of MPS that does not meet the American College of Rheumatology (ACR) diagnostic criteria for FM. No current injuries or integumentary abnormalities at the designated palpation sites.
3. FM group: Individuals who met the criteria for a diagnosis of FM based upon the ACR diagnostic criteria. No current injuries or integumentary abnormalities at the designated palpation sites.

Prior to testing, participants filled out a screening questionnaire with questions that represent the exclusion criteria which were used to determine ineligibility for this study. Participants who met the inclusion criteria and consented to participate were enrolled in the study. A California State University Dominguez Hills approved consent was read and signed by all participants prior to beginning data collection. Following consent, participant filled out a questionnaire to provide demographic information which included age, height, weight, arm dominance.

Following completion of the paperwork, all participants underwent testing from the primary investigator which was conducted between the hours of 8 am and 2pm. Participants were instructed to refrain from taking any related medication (e.g. pain medication) prior to testing. All participants underwent the same testing procedures and were blinded from the examiner's scores and other participants enrolled in the study.

For the reliability portion of the study, a total of 20 participants (10 MPS/FM and 10 control group) underwent 2 days of testing. Each testing session lasted approximately 45 minutes. After the reliability portion was complete, all other recruited subjects underwent 1 day of testing which lasted approximately 45 minutes.

The testing process consisted of 2-parts which were based upon the American College of Rheumatology (ACR) diagnostic criteria for FM. The protocol required the examiner to apply pressure to 18 pre-determined and 2 control points up to 4kg/cm2 at a rate of 1kg per second for a total of 4 seconds at each point, one time.12, 13 For Part I, the examiner applied a gradually increasing pressure using the thumb and digital pressure sensor at each pre-determined tender point. For Part II, the examiner applied a gradual increasing pressure using the algometer to the pre-determined tender points. For both Part I and II, the participant recorded their level of discomfort at each tender point using the MTPS and VAS pain scales once the examiner reached 4kg/cm2 of pressure or once a maximum level of pressure was felt. Participants were able to stop testing at any time. The examiner simultaneously recorded the patient's response using the PPTS scale for each tender point.

Collected data was transferred to SPSS v.22 (IBM SPSS, Chicago, IL). Means, standard error of mean (SEM), 95% confidence intervals (95% CI), and ranges of the descriptive data from each group was calculated. Group differences were calculated using the independent t-test. Six clinical questions were measured in this investigation which required specific parametric and non-parametric (ordinal data) statistical calculations. The P-value was considered significant at the .05 level using a two-tailed test (α2 =.05) for all clinical questions.

ELIGIBILITY:
Inclusion Criteria:

* Control group: Individuals with no current or prior diagnosis consistent with Myofascial Pain Syndrome (MPS) or Fibromyalgia (FM).
* MPS group: Individuals with a diagnosis of MPS that does not meet the American College of Rheumatology (ACR) diagnostic criteria for FM.
* FM group: Individuals who met the criteria for a diagnosis of FM based upon the ACR diagnostic criteria.

Exclusion Criteria:

* Current neurologic conditions (e.g. Multiple Sclerosis)
* Current metabolic conditions (e.g. Diabetic Neuropathy)
* Current systemic conditions (e.g. Rheumatoid Arthritis)
* Any skin or connective tissue problems (e.g. Marfan Syndrome)
* Current symptoms of numbness, tingling, burning, coldness, or pain in your back, hands, or feet.
* Any prior surgeries that may affect their ability to participate in this study.
* A pacemaker or electrical implant that may be affected by electronic equipment.
* Currently taking medications that may alter a subject's sensation or affect their ability to participate in this study.
* Current shingles or post-herpetic neuralgia.
* Current open skin wounds on your neck, arms, back, or legs
* Current injuries at the designated palpation sites.
* Currently having other medical conditions or limited function that might affect participation.
* The ability to tolerate testing duration and procedures.
* The ability to understand and complete all consent forms and questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups of participants were recruited for this study:
  * Control group: Individuals with no current or prior diagnosis consistent with Myofascial Pain Syndrome (MPS) or Fibromyalgia (FM).
  * MPS group: Individuals with a diagnosis of MPS that does not meet the American College of Rheumatology (ACR) diagnostic criteria for FM.
  * FM group: Individuals who met the criteria for a diagnosis of FM based upon the ACR diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold Scale | Baseline
  0-4 ordinal ranked scale (0-no pain to 4-intolerable pain)

SECONDARY OUTCOMES:
Visual Analog Pain Scale | Baseline
  Patient Related Outcome Measure for Pain
Manual Tender Point Survey (MTPS) | Baseline
  The MTPS is a version of the 11-point numeric pain rating scale for pain (ordinal scale)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Cheatham, DPT, PhD, Principal Investigator — CSUDH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ge HY, Wang Y, Danneskiold-Samsoe B, Graven-Nielsen T, Arendt-Nielsen L. The predetermined sites of examination for tender points in fibromyalgia syndrome are frequently associated with myofascial trigger points. J Pain. 2010 Jul;11(7):644-51. doi: 10.1016/j.jpain.2009.10.006. Epub 2009 Nov 14. PMID 19914876
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Alonso-Blanco C, Fernandez-de-las-Penas C, Morales-Cabezas M, Zarco-Moreno P, Ge HY, Florez-Garcia M. Multiple active myofascial trigger points reproduce the overall spontaneous pain pattern in women with fibromyalgia and are related to widespread mechanical hypersensitivity. Clin J Pain. 2011 Jun;27(5):405-13. doi: 10.1097/AJP.0b013e318210110a. PMID 21368661
- [Background] Alonso-Blanco C, Fernandez-de-Las-Penas C, de-la-Llave-Rincon AI, Zarco-Moreno P, Galan-Del-Rio F, Svensson P. Characteristics of referred muscle pain to the head from active trigger points in women with myofascial temporomandibular pain and fibromyalgia syndrome. J Headache Pain. 2012 Nov;13(8):625-37. doi: 10.1007/s10194-012-0477-y. Epub 2012 Aug 31. PMID 22935970
- [Background] Kothari SF, Kothari M, Zambra RF, Baad-Hansen L, Svensson P. Standardization of muscle palpation- methodological considerations. Clin J Pain. 2014 Feb;30(2):174-82. doi: 10.1097/AJP.0b013e31828c893d. PMID 24398392
- [Background] Sterling M. Pressure algometry: what does it really tell us? J Orthop Sports Phys Ther. 2011 Sep;41(9):623-4. doi: 10.2519/jospt.2011.0106. Epub 2011 Aug 31. No abstract available. PMID 21885903
- [Derived] Cheatham SW, Kolber MJ, Mokha GM, Hanney WJ. Concurrent validation of a pressure pain threshold scale for individuals with myofascial pain syndrome and fibromyalgia. J Man Manip Ther. 2018 Feb;26(1):25-35. doi: 10.1080/10669817.2017.1349592. Epub 2017 Jul 9. PMID 29456445